CLINICAL TRIAL: NCT07032818
Title: Communication Outreach for Navigation and Needs-based Care Transitions (CONNECT): A Pilot Randomized Controlled Trial
Brief Title: Adapted Hospital Discharge Intervention: the CONNECT Pilot
Acronym: CONNECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-45822; K23MD019068-01 (NIH)
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Communication Research
Keywords: Discharge instructions; Non-English language preference; Adapting hospital discharge

STUDY DESIGN:
Intervention Model Description: Two arm randomized controlled trial (2:1 intervention:control), Randomization stratified by language.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational intervention (Other): Participants randomized into this arm will receive current hospital discharge education and an additional post-discharge educational call.
  Interventions: Other: Additional post discharge phone call
- Standard of care (No Intervention): Participants randomized into this arm will receive current hospital discharge education.

INTERVENTIONS:
Other: Additional post discharge phone call — 24-72 hours after hospital discharge, a nurse will call participants to review the written After Visit Summary (AVS) given at discharge, including primary diagnosis, self-care instructions, emergency plan, medication changes, how and why to take medication, and scheduled follow up. These phone calls will take on average 10-15 minutes.
  Arms: Educational intervention

SUMMARY:
Hospital discharge is a dangerous time for patients: one in five will suffer an adverse event, such as a medication error, and nearly 25% will be readmitted within 30 days. This time is even more dangerous for patients with who face communication barriers, including those with non-English language preference (NELP), low health literacy, and the elderly.

The investigators will pilot a post-discharge educational intervention to reinforce written discharge instructions (known as the After Visit Summary or AVS) using a randomized controlled trial design (2:1 intervention: control). The control group will receive current standard of care discharge education which includes a nurse reviewing their AVS and an automated call in English that allows patients to numerically select types of problems/questions that are then escalated to a nurse who should return their call within a few days. The intervention group will receive the standard of care discharge education with the AVS and an additional post-discharge educational call delivered by a registered nurse or other qualified health professional with the option to have written instructions professionally translated and sent via MyChart message--if available in their preferred language.

ELIGIBILITY:
Inclusion Criteria:

* Registered language in Epic (written or spoken) is Spanish, Haitian Creole, Portuguese, Cape Verdean, or Vietnamese
* Admitted to medicine team at Boston Medical Center (BMC)
* Being discharged home (to the community)

Exclusion Criteria:

* On airborne infections precautions at time of recruitment
* On C diff precautions at time of recruitment
* On suicide precautions at time of recruitment
* Nurse report of participant displaying cognitive impairment, ongoing delirium, or aggression
* Discharge observed during a prior admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Retention success by linguistic group | 12 months
  Number of enrolled participants who completed all study assessments stratified by linguistic group.
Fidelity to the intervention | 12 months
  The number of scheduled educations calls that were completed for participants in the intervention arm based on nursing documentation in Epic.

SECONDARY OUTCOMES:
Acceptability of the intervention | 12 months
  The Acceptability of Intervention Measure (AIM) will be completed by participants in the intervention arm to assess acceptability. It has four questions with 5 Likert responses where 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree, The range of scores from 4 to 20 with higher scores indicating greater acceptability.
Feasibility of the intervention | 12 months
  Feasibility will be assessed by the number of participants in the intervention arm whose educational call was language concordant based on nursing documentation in Epic.
Patient Understanding of Discharge Instruction (UDI) Scale | 12 months
  Assessed by a composite score of six key domains of discharge instructions (primary diagnosis, self-care instructions, return precautions, medication changes, medication indications, follow-up) as determined by physician adjudicators (1=poor, 4 = near perfect). Higher scores demonstrate better understanding.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Austad, MD MPH, Principal Investigator — Boston Medical Center, Family Medicine
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No